CLINICAL TRIAL: NCT02745262
Title: Retrospective Cohort Study of Overall Survival and Disease-free Survival in Breast Cancer Patients Who Underwent Controlled Ovarian Stimulation (COS)
Brief Title: Overall Survival and Disease-free Survival in Breast Cancer Patients Under COS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IVI Vigo (Other)
Responsible Party: Sponsor
Other Study IDs: 1405-VIG-030-EM
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Controlled ovarian stimulation: No drugs are administered. It is an observational study. Collect retrospectively the follow-up data
  Interventions: Other: Collect retrospectively the follow-up data
- Non Controlled ovarian stimulation: No drugs are administered. It is an observational study. Collect retrospectively the follow-up data
  Interventions: Other: Collect retrospectively the follow-up data

INTERVENTIONS:
Other: Collect retrospectively the follow-up data — Collect retrospectively the follow-up data. Each patient is called in order to request data authorization, to complete and track information.

SUMMARY:
The main objective of the study is to evaluate the overall survival and disease-free survival in breast cancer patients under 40 years old. They underwent controlled ovarian stimulation (COS) for fertility preservation versus women of the same age, type and stage of breast cancer, who have not been subjected to COS.

DETAILED DESCRIPTION:
Breast cancer is a disease where the tumor size, lymph node involvement and histological grade provide rich information about prognosis and enable to stage the disease. As in any other oncological pathology, stage of disease at diagnosis is the major determining factor for estimating survival. Ovarian stimulation for fertility preservation is performed in this study, in patients with stage I-II (TNM) after the neoplasia is treated (surgical removal of the tumor) prior to systemic therapy, when indicated.

Among young women there is a greater incidence of basal type tumors and HER2 (human epidermal growth factor receptor 2), which do not always express hormone receptors. In early stages of the disease, the controlled ovarian stimulation procedure, after removal of the tumor, has not revealed any worsening in the prognosis of the disease, in terms of overall survival and disease-free survival (absence of local or distant recurrence).

It is a study that aims to collect data retrospectively from 2008 to 31 December 2015. To this end, we will collect the follow-up data, up to 5 years for patients from 2008, 2009 and 2010. Four years for patients in 2011, 3 years for 2012, 2 years for 2013, one year for those included until 31 December 2014 and patients followed until 31 December 2015. Each patient is called in order to request data authorization, to complete and track information.

ELIGIBILITY:
Inclusion Criteria:

* Age under 40 years ( at the time of diagnosis)
* TNM stage I- II
* Authorization of the fertility preservation multidisciplinary committee

Exclusion Criteria:

* Contraindications for pregnancy
* previous history of infertility
* Previous history of ovarian surgery
* Prior chemotherapy
* History of pelvic radiation
* Diabetes Mellitus
* Hypertension
* renal failure
* liver failure
* autoimmune disease.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Age under 40 years ( at the time of diagnosis) TNM stage I- II Authorization of the fertility preservation multidisciplinary committee
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival rate | Up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Principal Investigator — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cobo A, Garcia-Velasco JA, Domingo J, Remohi J, Pellicer A. Is vitrification of oocytes useful for fertility preservation for age-related fertility decline and in cancer patients? Fertil Steril. 2013 May;99(6):1485-95. doi: 10.1016/j.fertnstert.2013.02.050. Epub 2013 Mar 29. PMID 23541405
- [Result] Oktay K, Rodriguez-Wallberg K, Munster P. Ovarian protection during adjuvant chemotherapy. N Engl J Med. 2015 Jun 4;372(23):2268-9. doi: 10.1056/NEJMc1504241. No abstract available. PMID 26039611
- [Result] Frydman R, Grynberg M. Introduction: Female fertility preservation: innovations and questions. Fertil Steril. 2016 Jan;105(1):4-5. doi: 10.1016/j.fertnstert.2015.10.035. Epub 2015 Nov 21. PMID 26612064